CLINICAL TRIAL: NCT00001571
Title: A Pilot Study of Non-Hodgkin's Lymphoma: Chemotherapy and Blood Levels of Organochlorines
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970075; 97-C-0075
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: HIV Infections; Lymphoma, AIDS-Related; Lymphoma, Non-Hodgkin
Keywords: Cancer; DDT, PCB; Epidemiology; Pesticides; Serum
MeSH Terms: conditions — HIV Infections; Lymphoma, AIDS-Related; Lymphoma, Non-Hodgkin; Neoplasms

SUMMARY:
Non-Hodgkin's lymphoma (NHL) is the third most rapidly increasing cancer in the United States. HIV-related NHL is responsible for some of the increase since the early 1980s. However, it cannot explain the steady increase in the incidence rates in earlier years, nor the entire increase shown recently. A possible role of environmental exposures is receiving attention. One possibility is that exposure to organochlorines (OCs) may be related to the occurrence of NHL. NCI is currently designing a large population-based case-control study to investigate this hypothesis further by analyzing OC levels in blood collected at the time of interview from cases of NHL and their matched controls. At the time of these interviews, cases in the main case-control study would most likely have already received chemotherapy. If chemotherapy changes the blood levels of OCs, this may lead to misclassification of exposure among cases and eventually to biased risk estimates. The purpose of this pilot study is to estimate the bias due to measuring the serum levels of OCs in cases during or after chemotherapy. Twenty newly diagnosed patients will be recruited for the study. From each patient, four consecutive blood samples, one prior to, two during, and one after chemotherapy, will be collected. Forty pairs of pre-existing cryopreserved serum samples (pre- and post-treatment) taken from the NHL patients who participated in an earlier NCI clinical study will also be included in this study. Samples will be assayed for OC levels. The results will be used to plan and to interpret another large case-control study (the main study).

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma (NHL) is the third most rapidly increasing cancer in the United States. HIV-related NHL is responsible for some of the increase since the early 1980s. However, it cannot explain the steady increase in the incidence rates in earlier years, nor the entire increase shown recently. A possible role of environmental exposures is receiving attention. One possibility is that exposure to organochlorines (OCs) may be related to the occurrence of NHL. NCI is currently designing a large population-based case-control study to investigate this hypothesis further by analyzing OC levels in blood collected at the time of interview from cases of NHL and their matched controls. At the time of these interviews, cases in the main case-control study would most likely have already received chemotherapy. If chemotherapy changes the blood levels of OCs, this may lead to misclassification of exposure among cases and eventually to biased risk estimates. The purpose of this pilot study is to estimate the bias due to measuring the serum levels of OCs in cases during or after chemotherapy. Twenty newly diagnosed patients will be recruited for the study. From each patient, four consecutive blood samples, one prior to, two during, and one after chemotherapy, will be collected. Forty pairs of pre-existing cryopreserved serum samples (pre- and post-treatment) taken from the NHL patients who participated in an earlier NCI clinical study will also be included in this study. Samples will be assayed for OC levels. The results will be used to plan and to interpret another large case-control study (the main study).

ELIGIBILITY:
All NHL patients who have not previously received chemotherapy and who are admitted to the NCI Clinical Center to be enrolled in trails will be eligible for the study.

All histological subtypes and stages.

Any NHL patient who is between the ages of 20 and 74.

Must be able to give informed consent.

No NHL patient HIV positive will be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1997-02; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cantor KP, Blair A, Everett G, Gibson R, Burmeister LF, Brown LM, Schuman L, Dick FR. Pesticides and other agricultural risk factors for non-Hodgkin's lymphoma among men in Iowa and Minnesota. Cancer Res. 1992 May 1;52(9):2447-55. PMID 1568215
- [Background] Gammon MD, Wolff MS, Neugut AI, Terry MB, Britton JA, Greenebaum E, Hibshoosh H, Levin B, Wang Q, Santella RM. Treatment for breast cancer and blood levels of chlorinated hydrocarbons. Cancer Epidemiol Biomarkers Prev. 1996 Jun;5(6):467-71. PMID 8781744
- [Background] Hoffman W. Organochlorine compounds: Risk of non-Hodgkin's lymphoma and breast cancer? Arch Environ Health. 1996 May-Jun;51(3):189-92. doi: 10.1080/00039896.1996.9936015. PMID 8687239